CLINICAL TRIAL: NCT01933074
Title: Clinical and Biochemical Evidence of Neurogenic Inflammation in Women With Urinary Urgency
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 817047
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2013-01

CONDITIONS: Overactive Bladder
Keywords: Urinary Urgency
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — First morning urine specimens are collected from each subject after completing questionnaires - one week from initial visit or at follow-up visit.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to gain a better understanding of what causes urinary urgency in women by asking about different symptoms and measuring biomarker levels in their urine. Understanding the underlying causes of urinary urgency will allow us to develop treatment options to better take care of women with urinary urgency.

DETAILED DESCRIPTION:
We propose to test the hypothesis that urinary urgency in women is caused by neurogenic inflammation that is manifested clinically as neuropathic pain and associated with the expression of neuroinflammatory biomarkers in the urine.

ELIGIBILITY:
Inclusion criteria: Age > 18, urinary urgency (at least mild bother on a single item Urgency Scale), and negative urine dipstick on clean catch.

-

Exclusion Criteria:: Urinary incontinence (greater than mild on the Incontinence Severity Index), recent (<6week) urinary tract infection, active or recent(<3month) nephrolithiasis, prior diagnosis of congenital urinary tract abnormality, known neurological disorder (multiple sclerosis, Parkinson's, spina bifid, spinal cord injury), recent pregnancy < 3 months, prior sacral nerve stimulation or Botox injection.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urogynecology clinic
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To determine the association between the severity of neuropathic pain and the severity of urinary symptoms in women with urinary urgency. | 1 year
  We propose a prospective cross-sectional study. We will recruit 137 women with urinary urgency and without incontinence or infection. All women will complete validated symptom questionnaires to measure neuropathic pain, urinary, bowel, sexual symptoms and quality of life. All patients will bring a first morning clean catch urine void to the office on ice within one week of completing the questionnaires. The specimen will be transported to the lab within 24 hours and stored at -80 degrees. Enzyme-linked immunosorbent assays (ELISA) will be used to determine expression of urinary creatinine and neuropeptides. The primary outcome will be the severity of urinary symptoms as measured by the Interstitial Cystitis Symptom Index.

SECONDARY OUTCOMES:
The association between neuropathic pain and the expression of potential neural biomarkers in the urine of women with urinary urgency. | 1 year
  To determine the association between the severity of neuropathic pain and expression of urinary neurotrophic peptides in women with urgency. We hypothesize that in women with urinary urgency, increasing severity of neuropathic pain will be associated with increasing levels of urinary neurotrophic peptides NGF and BDNF. Nerve growth factor (NGF) and Brain-Derived Neurotrophic factor (BDNF) - NGF and BDNF are neurotrophic growth factors that are released in urine from different cell types in the bladder wall making urine a convenient sample for measurement of their levels. Activation of the myelinated A fiber and unmyelinated C fibers in the bladder wall can lead to an elevation in NGF and BDNF levels, sensitization of bladder afferent pathways and development of neurogenic inflammation in the urinary bladder [2,3].

CONTACTS AND LOCATIONS:
Overall Officials: Uduak Umoh-Andy, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Pelvic and Sexual Health Insitute, Philadelphia, Pennsylvania, United States